CLINICAL TRIAL: NCT03760510
Title: The Effect of Adhesive Versus Endotracheal Tube Fastener in Critically Ill Adults: The Endotracheal Tube Securement Study
Brief Title: Endotracheal Tube Securement Study
Acronym: ETTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Todd Rice, Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB #170596
Record Dates: First submitted 2018-11-26; First posted 2018-11-30 (Actual); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Mechanical Ventilation Complication
Keywords: endotracheal tube; tube fastener; facial skin tear; lip ulcer; endotracheal tube dislodgement
MeSH Terms: interventions — Surgical Tape

STUDY DESIGN:
Intervention Model Description: The endotracheal tube securement study was a pragmatic, single center, open-label, randomized trial comparing the effect of adhesive tape versus endotracheal tube fastener (Hollister AnchorFast Guard) among critically ill adults requiring intubation and mechanical ventilation for at least 24 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Adhesive Tape (Experimental): Patients in adhesive tape arm had endotracheal tube secured with adhesive tape
  Interventions: Device: Adhesive Tape
- Tube Fastener (Experimental): Patients in the tube fastener arm had endotrachel tube secured with tube fastener
  Interventions: Device: Tube Fastener

INTERVENTIONS:
Device: Tube Fastener — Endotrachel tube secured with tube fastener
  Other Names: Hollister AnchorFast
  Arms: Tube Fastener
Device: Adhesive Tape — Endotracheal tube secured with adhesive tape.
  Arms: Adhesive Tape

SUMMARY:
To evaluate the safety and efficacy of endotracheal tube securement techniques, a pragmatic, randomized controlled trial will compare the effect of adhesive tape versus endotracheal tube fastener on complications including lip ulcers, facial skin tears, endotracheal tube dislodgement, and ventilator associated pneumonia among critically ill adults requiring intubation and mechanical ventilation for at least 24 hours.

DETAILED DESCRIPTION:
Background: The optimal securement method of endotracheal tubes is unknown, but should provide adequate security while minimizing complications. This study tests the hypothesis that use of an endotracheal tube fastener would reduce complications among critically ill adults undergoing endotracheal intubation. This hypothesis will be tested in a pragmatic, single center, randomized trial comparing the effect of adhesive tape versus endotracheal tube fastener (Hollister) among critically ill adults requiring intubation and mechanical ventilation for at least 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patient intubated prior to admission to the MICU and the intubation time was less than 12 hours from the time of admission
* Patients intubated in the MICU for greater than 24 hours

Exclusion Criteria:

* intubated greater than 12 hours prior to admission to the MICU
* presence of oral mucosa or facial skin breakdown prior to enrollment
* required nasotracheal intubation,
* had a documented allergy to tape
* pregnant
* prisoners

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-04-14 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janna Landsperger, ACNP, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
publication in a peer-reviewed medical journal

REFERENCES:
- [Derived] Landsperger JS, Byram JM, Lloyd BD, Rice TW; Pragmatic Critical Care Research Group. The effect of adhesive tape versus endotracheal tube fastener in critically ill adults: the endotracheal tube securement (ETTS) randomized controlled trial. Crit Care. 2019 May 7;23(1):161. doi: 10.1186/s13054-019-2440-7. PMID 31064406

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adhesive Tape | Tube Fastener
Started | 250 | 250
Completed | 145 | 153
Not Completed | 105 | 97
Not completed — Not ventilated for 24 hours | 105 | 97

BASELINE CHARACTERISTICS:
Population: Eligible patients had to be intubated for at least 24 hours.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adhesive Tape | Tube Fastener | Total
Number analyzed (Participants) | 145 | 153 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (16.1) | 53.2 (16.4) | 55.8 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 76 | 142
  Male | 79 | 77 | 156
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 19 | 42
  White | 111 | 122 | 233
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 12 | 23
APACHE II [Mean (Standard Deviation); unit: units on a scale] — Severity of Illness Score. Scores range from minimum value of 0 to maximum value of 71 points. Higher score indicates greater severity of illness.
  units on a scale | 27.4 (8.7) | 26.0 (8.9) | 26.7 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Any Incidence of the Following: Presence of Lip Ulcer, Endotracheal Tube Dislodgement, or Facial Skin Tears From the Time of Randomization to the Earlier of Death or 48 Hours After Extubation
Description: Rate per 1000 ventilator days of any incidence of the following: presence of lip ulcer, endotracheal tube dislodgement, or facial skin tears from the time of randomization to the earlier of death or 48 hours after extubation
Time Frame: 48 hours post extubation up to 3 months
Population: Enrolled patients ventilated for at least 24 hours who had primary outcome data
Measure: Mean (95% Confidence Interval); unit: events per 1000 ventilator days
Arm/Group | Adhesive Tape | Tube Fastener
Number analyzed (Participants) | 145 | 153
events per 1000 ventilator days | 52.6 [47.4 to 57.8] | 22.0 [16.3 to 27.7]

2. Secondary Outcome: Number of Participants With Lip Ulcers
Description: Presence of lip ulcer
Time Frame: 48 hours post extubation up to 3 months
Population: Enrolled patients mechanically ventilated for at least 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Adhesive Tape | Tube Fastener
Number analyzed (Participants) | 145 | 153
Participants | 11 | 4

3. Secondary Outcome: Number of Participants With Facial Skin Tear
Description: presence of facial skin tear
Time Frame: 48 hours post extubation up to 3 months
Population: Enrolled participants receiving mechanical ventilation for at least 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Adhesive Tape | Tube Fastener
Number analyzed (Participants) | 145 | 153
Participants | 3 | 2

4. Secondary Outcome: Number of Participants With Ett Dislodgement
Description: frequency of ett dislodgement
Time Frame: duration of intubation up to 3 months
Population: Enrolled participants receiving mechanical ventilation for at least 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Adhesive Tape | Tube Fastener
Number analyzed (Participants) | 145 | 153
Participants | 15 | 6

ADVERSE EVENTS:
Time Frame: Until 48 hours after extubation
Description: Adverse events were collected prospectively and included self-extubations.
Arm/Group | Adhesive Tape | Tube Fastener
All-Cause Mortality (participants affected / at risk) | 54/145 | 57/153
Serious Adverse Events (participants affected / at risk) | 2/145 | 2/153
Other Adverse Events (participants affected / at risk) | 0/145 | 0/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adhesive Tape (N=145) | Tube Fastener (N=153)
Self-Extubation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) — Patient self-extubation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT03760510/Prot_SAP_000.pdf